CLINICAL TRIAL: NCT05132322
Title: Eliminating Monitor Overuse (EMO) Hybrid Effectiveness-Deimplementation Trial
Brief Title: Eliminating Monitor Overuse Trial (EMO Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Pennsylvania (Other); Boston Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Pediatric Research in Inpatient Settings (PRIS) Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-018560; U01HL159880 (NIH)
Record Dates: First submitted 2021-11-10; First posted 2021-11-24 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Bronchiolitis Acute Viral
Keywords: pulse oximetry; deimplementation; cluster-randomized trial; effectiveness-implementation hybrid trial; implementation science

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unlearning Only (Active Comparator): Includes educational outreach and audit & feedback.
  Interventions: Behavioral: Educational Outreach; Behavioral: Audit & Feedback (unit level); Behavioral: Audit & Feedback (real time, individual-level)
- Unlearning + Substitution (Experimental): Includes educational outreach, audit & feedback, and an electronic health record-integrated clinical pathway to support appropriate use of pulse oximetry.
  Interventions: Behavioral: Educational Outreach; Behavioral: Audit & Feedback (unit level); Behavioral: Audit & Feedback (real time, individual-level); Behavioral: Clinical Pathway Integrated into Electronic Health Record

INTERVENTIONS:
Behavioral: Educational Outreach — Educational outreach includes staff-targeted educational materials and outreach sessions summarizing the current evidence and guideline recommendations for pulse oximetry use in bronchiolitis.
Behavioral: Audit & Feedback (unit level) — Weekly unit-level feedback of each hospital's guideline-concordant practice will be distributed to sites in the form of a visual dashboard that includes comparisons over time and between hospitals. The dashboard will then be shared locally on a weekly basis with clinicians in person and electronically.
Behavioral: Audit & Feedback (real time, individual-level) — Real-time feedback will occur at the individual clinician level. When collecting data on an individual patient, data collectors encountering guideline-discordant continuous monitoring are empowered to briefly ask any available clinician responsible for that patient's care, in a nonjudgmental way, about indications for monitoring that patient. The clinician is ultimately responsible for deciding if any changes are indicated.
Behavioral: Clinical Pathway Integrated into Electronic Health Record — Clinical pathways guide clinicians step-by-step through evidence-based care. Based on the existing guidelines for physiologic monitoring in bronchiolitis, the pathway will clearly specify (a) situations when it is appropriate to initiate intermittent SpO2 measurement instead of continuous SpO2 monitoring, and (b) when it is appropriate to discontinue continuous SpO2 monitoring altogether, and transition to intermittent SpO2 measurement. In order to be visible to clinicians as they perform patient care, the pathway will be integrated into the electronic health record at sites randomized to this intervention.
  Arms: Unlearning + Substitution

SUMMARY:
The purpose of this study is to identify the optimal deimplementation strategies for an overused practice: continuous pulse oximetry monitoring of children hospitalized with bronchiolitis who are not receiving supplemental oxygen.

ELIGIBILITY:
Population 1a: Hospital staff who complete study questionnaires.

Inclusion Criteria:

* Nurse or physician fluent in English and employed full-time by the hospital, affiliated practice, or affiliated university who cared for bronchiolitis patients on a unit participating in the trial during at least 5 days of the most recent bronchiolitis season
* Hospital administrator fluent in English who oversaw the care of bronchiolitis on a local level (e.g. nurse manager) or a hospital level (e.g. Chief Quality and Safety Officer)

Exclusion Criteria:

• Under the direct supervision of study or site principal investigator(s)

Population 1b: Hospital staff who participate in qualitative interviews

In Aim 2, we will conduct semi-structured interviews with physicians and nurses who provide care to bronchiolitis patients in participating units at the 5 hospitals with the highest and 3 hospitals with the lowest sustainability (8 hospitals total; up to maximum of 8 interviews/hospital). Maximum anticipated enrollment 64.

Inclusion criteria:

* Nurses or Physicians who cared for bronchiolitis patients on a unit participating in the trial during at least 5 days of the most recent bronchiolitis season
* Employed full-time by the hospital, affiliated practice, or affiliated university
* Fluent in English

Exclusion criteria:

• No exclusion criteria

Population 2a: Bronchiolitis patients directly observed while not receiving supplemental oxygen ("in room air," for primary trial outcome)

Inclusion Criteria:

* Infants and children 2 months through 23 months old
* Hospitalized on non-ICU wards participating in the trial
* Cared for by generalist inpatient services (e.g. general pediatrics, hospital medicine)
* Primary diagnosis of bronchiolitis in most recent physician progress note
* Not actively receiving supplemental oxygen ("in room air")
* Last documented receipt of supplemental oxygen >1 hour prior to direct observational data collection

Exclusion Criteria:

* Documented apnea or cyanosis during the current illness
* Extreme prematurity (<28 weeks completed gestation)
* Cardiac disease
* Pulmonary hypertension
* Chronic lung disease
* Home oxygen requirement
* Neuromuscular disease
* Immunodeficiency
* Cancer
* Severe Acute Respiratory Syndrome Coronavirus 2 (Covid-19 / SARS-CoV-2)-related illness (known or suspected, including multisystem inflammatory syndrome in children multi-system inflammatory syndrome in children (MIS-C)

Population 2b: Bronchiolitis patients directly observed while receiving supplemental oxygen (for underuse evaluation).

Inclusion Criteria:

* Infants and children 2 months through 23 months old
* Hospitalized on non-ICU wards participating in the trial
* Cared for by generalist inpatient services (e.g. general pediatrics, hospital medicine)
* Primary diagnosis of bronchiolitis in most recent physician progress note
* Actively receiving ≥2 Liters/minute (2L/min) supplemental oxygen or 21% room air flow

Exclusion Criteria:

* Extreme prematurity (<28 weeks completed gestation)
* Cardiac disease
* Pulmonary hypertension
* Chronic lung disease
* Home oxygen requirement
* Neuromuscular disease
* Immunodeficiency
* Cancer
* Severe Acute Respiratory Syndrome Coronavirus 2 [Covid-19 / SARS-CoV-2 (known or suspected)]

Population 3: Parents or guardians of bronchiolitis patients who participate in qualitative interviews.

Inclusion Criteria:

* Their child was hospitalized for bronchiolitis on a unit participating in the trial during the most recent bronchiolitis season
* Their child was found to be in room air during Aim 1 data collection
* Fluent in English

Exclusion criteria:

• They are an employee of the hospital or a hospital volunteer

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32357 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sustainability of guideline-concordant deimplementation of continuous pulse oximetry monitoring | 3 years
  Sustainability of guideline-concordant deimplementation of continuous pulse oximetry (SpO2) monitoring is the primary trial outcome. It is calculated based on penetration (outcome 2). Sustainability will be measured longitudinally based on calculating the differences in the penetration of guideline-concordant practice at baseline, compared to the penetration during the sustainability phase.

SECONDARY OUTCOMES:
Penetration | Up to 4 years
  Penetration is calculated as the percentage of bronchiolitis patients who are in room air (not receiving any supplemental oxygen) and are receiving guideline-concordant care (this means they are not being continuously SpO2-monitored). The continuous monitoring status is determined using direct observation on hospital units.
Acceptability of deimplementation | Up to 3 years
  Acceptability of deimplementation among staff measured by questionnaire. Items are adapted from the validated Acceptability of Implementation Measure (AIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better acceptability. The items are analyzed individually and not summed to a total score.
Feasibility of deimplementation | Up to 3 years
  Feasibility of deimplementation among staff measured by questionnaire. Items are adapted from the validated Feasibility of Implementation Measure (FIM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better feasibility. The items are analyzed individually and not summed to a total score.
Appropriateness of deimplementation | Up to 3 years
  Appropriateness of deimplementation among staff measured by questionnaire. Items are adapted from the validated Implementation Appropriateness Measure (IAM) and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better appropriateness. The items are analyzed individually and not summed to a total score.
Perceived safety of deimplementation | Up to 3 years
  Perceived safety of deimplementation among staff measured by questionnaire. Items are adapted from those used in the pilot study preceding this trial and are rated on a 5-point Likert scale ranging from 1 to 5, with 1 indicating "Completely disagree" and 5 indicating "Completely agree." Higher scores indicate better agreement with each question.
Cost of deimplementation strategies | Up to 3 years
  Cost of delivering each of the strategies will be assessed using a pragmatic Time-Driven Activity Based Costing method developed specifically for economic analysis of implementation strategies.
Length of Hospital Stay | Up to 4 years
  The length of hospital stay is the duration of time that elapses between the time a patient is admitted with bronchiolitis to an inpatient unit of the hospital until the time they are discharged from the hospital, using data manually abstracted from the electronic health record chart.
Duration of Oxygen Supplementation | Up to 4 years
  The oxygen supplementation duration is the total duration of time during which a patient is documented as receiving supplemental oxygen during hospitalization.

OTHER OUTCOMES:
Exploratory long-term sustainability | 4 years
  Exploratory long-term sustainability is calculated based on penetration. Penetration is the percentage of bronchiolitis patients who are in room air (not receiving any supplemental oxygen) and are receiving guideline-concordant care (this means they are not being continuously SpO2-monitored). The continuous monitoring status is determined using direct observation on hospital units.
  In this exploratory outcome investigators are using an alternative definition of sustainability in which, in order to meet criteria for having successfully sustained a practice change, hospitals must first (a) experience a significant increase in penetration between baseline and active deimplementation, and then (b) maintain the increased penetration at ≥90% of the active deimplementation phase level through the end of the sustainability period.
Routinization of guideline-concordant deimplementation | Up to 3 years
  Routinization is a dimension of the Slaghuis Measurement Instrument for Sustainability of Work Practices. Routinization is the process in which clinicians develop new routines such that the intended practice changes become part of their everyday work.
Institutionalization of guideline-concordant deimplementation | Up to 3 years
  Institutionalization is a dimension of the Slaghuis Measurement Instrument for Sustainability of Work Practices. Institutionalization is the process in which the organization embeds the intended practice change into its existing systems and structures.
Implementation Climate | Up to 3 years
  Implementation Climate is whether the environment expects, supports, and rewards deimplementation of continuous SpO2 monitoring. Investigators will measure Implementation Climate using items from the Implementation Climate Scale. This is an 18-item scale with each item having 5 response options from 0 through 4. Higher total scores indicate better implementation climate.
Implementation Leadership | Up to 3 years
  Implementation Leadership is leader behaviors that include being proactive, knowledgeable, supportive, and persevering around deimplementation of continuous SpO2 monitoring. Implementation Leadership will be measured using items from the Implementation Leadership Scale. This is a 12-item scale with each item having 5 response options from 0 through 4. Higher total scores indicate better implementation leadership.
Psychological reactance | Up to 3 years
  Assessment of psychological reactance by questionnaire will be performed using validated items from seminal research in psychological reactance in health communication. This includes dimensions of freedom threat, emotional response, and cognitive response to deimplementation. Items are rated on 5-point Likert scales ranging from 0 through 4 with higher scores indicating more reactance for some items, and less reactance on other items. The items are analyzed individually and not summed to a total score.
Underuse of Pulse Oximetry Monitoring in High Risk Patients | Up to 4 years
  Underuse is defined as failing to continuously SpO2 -monitor bronchiolitis patients receiving
  ≥2L/min supplemental oxygen (a marker of more severe disease). It is calculated as the percentage of bronchiolitis patients who are receiving ≥2L/min supplemental oxygen, and are not being continuously SpO2-monitored. It is measured using direct observation.
Number of Bronchiolitis Patients with Emergency Hypoxemic Events | Up to 4 years
  Investigators will collect data on emergency events occurring in bronchiolitis patients as a potential unintended consequence of deimplementation efforts. Investigators will identify code blue and rapid response team activations in bronchiolitis patients who were unmonitored at the time of the event and were subsequently found to be hypoxemic to <85% at the time of the event when SpO2 monitors were applied. These outcomes will be extracted from local patient safety databases (e.g., local rapid response team activation logs).
Number of Bronchiolitis Patients with Readmissions Featuring Hypoxemia Upon Re-Presentation | Up to 4 years
  Investigators will collect data on readmissions occurring in bronchiolitis patients as a potential unintended consequence of deimplementation efforts. Investigators will identify readmissions of bronchiolitis patients to the hospital within 7 days of discharge who were found to be hypoxemic to <85% upon re-presentation to the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Bonafide, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia; Rinad S Beidas, PhD, Principal Investigator — Northwestern University
Locations (58):
- United States (57):
  - Children's of Alabama, Birmingham, Alabama
  - Banner University Medical Center- Diamond Children's, Tucson, Arizona
  - University of California Davis, Davis, California
  - Rady Children's Hospital/UCSD, Encinitas, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Children's Hospital at Dartmouth-Hitchcock, Lebanon, New Hampshire
  - CHOP Pediatric Care at Penn Medicine/Princeton Health, Princeton, New Jersey
  - CHOP Care Network at Virtua, Voorhees Township, New Jersey
  - Albany Medical Center, Albany, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - NYP-Morgan Stanley Children's Hospital, New York, New York
  - Komansky Children's Hospital/New York Presbyterian Medical Center /Weill Cornell Medicine, New York, New York
  - University of Rochester Golisano Children's Hospital, Rochester, New York
  - Upstate Golisano Children's Hospital, Syracuse, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - CHOP King of Prussia Hospital, King of Prussia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Reading Hospital, Tower Health, Reading, Pennsylvania
  - CHOP Grand View Hospital, Sellersville, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Children's Memorial Hermann, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Texas Children's Hospital West Campus, Houston, Texas
  - Texas Children's Hospital The Woodlands, The Woodlands, Texas
  - Utah Valley Hospital, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont Children's Hospital, Burlington, Vermont
  - Inova Children's Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Hoops Family Children's Hospital at Marshall University, Huntington, West Virginia
  - Children's Wisconsin, Milwaukee, Wisconsin
- Alberta Children's Hospital, Calgary, Canada

REFERENCES:
- [Derived] Xiao R, Bonafide CP, Williams NJ, Cidav Z, Landrigan CP, Faerber J, Makeneni S, Wolk CB, Schondelmeyer AC, Brady PW, Beidas RS, Schisterman EF. Eliminating Monitor Overuse (EMO) type III effectiveness-deimplementation cluster-randomized trial: Statistical analysis plan. Contemp Clin Trials Commun. 2023 Oct 2;36:101219. doi: 10.1016/j.conctc.2023.101219. eCollection 2023 Dec. PMID 37842322
- [Derived] Faerber JA, Xiao R, Makeneni S, Schisterman EF, Brady PW, Schondelmeyer AC, Landrigan CP, Lucey K, Lee V, Gregory PF, Prasto J, Parthasarathy P, Greenfield M, Solomon C, Brent CR, Albanowski K, Beidas RS, Bonafide CP; Pediatric Research in Inpatient Settings (PRIS) Network. Sustainment of continuous pulse oximetry deimplementation: Analysis of Eliminating Monitor Overuse study data from six hospitals. J Hosp Med. 2023 Aug;18(8):724-729. doi: 10.1002/jhm.13154. Epub 2023 Jun 28. PMID 37380625
- [Derived] Bonafide CP, Xiao R, Schondelmeyer AC, Pettit AR, Brady PW, Landrigan CP, Wolk CB, Cidav Z, Ruppel H, Muthu N, Williams NJ, Schisterman E, Brent CR, Albanowski K, Beidas RS; Pediatric Research in Inpatient Settings (PRIS) Network. Sustainable deimplementation of continuous pulse oximetry monitoring in children hospitalized with bronchiolitis: study protocol for the Eliminating Monitor Overuse (EMO) type III effectiveness-deimplementation cluster-randomized trial. Implement Sci. 2022 Oct 21;17(1):72. doi: 10.1186/s13012-022-01246-z. PMID 36271399